CLINICAL TRIAL: NCT06132009
Title: Predictive Value of Preoperative Evaluation in Cases of Recurrent Endometriosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Evrim Ebru Kovalak, Medical Doctor, gynecologist, Bagcilar Training and Research Hospital
Other Study IDs: 2023/05/11/030
Record Dates: First submitted 2023-11-07; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Endometriosis
Keywords: Endometriosis; prevention & control; preoperative procedures
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Remission group: Group of women who underwent cystectomy or unilateral oophorectomy due to endometriosis but were in remission during follow-up
  Interventions: Procedure: Surgery of endometriosis
- Recurrent group: Group of women who underwent cystectomy or unilateral oophorectomy due to endometriosis but developed an endometrioma of at least 2 cm in size in a single ovary during follow-up.
  Interventions: Procedure: Surgery of endometriosis

INTERVENTIONS:
Procedure: Surgery of endometriosis — Cystectomy or unilateral oophorectomy due to endometriosis

SUMMARY:
To investigate the effect of preoperative evaluation parameters in predicting recurrent disease in women who have undergone cystectomy or unilateral salpingo-oophorectomy due to endometriosis.

DETAILED DESCRIPTION:
Endometriosis is an estrogen-dependent gynecological disease characterized by the presence of endometrial-like tissue outside the uterine cavity, associated with pelvic pain and subfertility. Despite its benign character, endometriosis can recur after surgery and continues to be a disease that disrupts the quality of life of millions of women. This study aimed to examine the risk factors in women who underwent cystectomy or unilateral salpingo-oophorectomy due to endometriosis but had a recurrence. Therefore, the predictive value of parameters such as preoperative biochemical parameters, cyst size and the revised American Society for Reproductive Medicine (rASRM) Scoring system will be examined in recurrent cases.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-50 who had a cystectomy or unilateral oophorectomy due to endometriosis

Exclusion Criteria:

* Women who have had bilateral oophorectomy due to endometriosis
* Malignant conditions
* Smoking
* Women with autoimmune disease

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: All women between the ages of 18-50 who were followed up in our clinic after cystectomy or unilateral oophorectomy due to endometriosis.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Prediction of endometriosis recurrence | 6-180 months
  Which women are more likely to have recurrence after endometriosis surgery?

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Ebru Kovalak, MD, Principal Investigator — Bagcilar Training and Research Hospital
Locations (1):
- Bagcilar Teaching and Research Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hidari T, Hirata T, Arakawa T, Koga K, Neriishi K, Fukuda S, Nakazawa A, Nagashima N, Ma S, Sun H, Takamura M, Harada M, Hirota Y, Wada-Hiraike O, Fujii T, Osuga Y. Contralateral ovarian endometrioma recurrence after unilateral salpingo-oophorectomy. BMC Womens Health. 2019 May 2;19(1):59. doi: 10.1186/s12905-019-0760-z. PMID 31046768
- See also: Hidari T, Hirata T, Arakawa T, Koga K, Neriishi K, Fukuda S, Nakazawa A, Nagashima N, Ma S, Sun H, Takamura M, Harada M, Hirota Y, Wada-Hiraike O, Fujii T, Osuga Y. Contralateral ovarian endometrioma recurrence after unilateral salpingo-oophorectomy. — https://doi.org/10.1186/s12905-019-0760-z

DOCUMENTS (1):
  • Informed Consent Form (2019-12-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT06132009/ICF_000.pdf